CLINICAL TRIAL: NCT04831515
Title: Performance Evaluation of Two Daily Disposable Toric Lens Designs in Habitual Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-122
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A (Experimental): daily disposable soft contact lens - test lens
  Subjects will be randomized to wear test lenses for one week and then cross-over to control lenses for one week.
  Interventions: Device: Lens A; Device: Lens B
- Lens B (Active Comparator): daily disposable soft contact lens - control lens
  Subjects will be randomized to wear control lenses for one week and then cross-over to test lenses for one week.
  Interventions: Device: Lens A; Device: Lens B

INTERVENTIONS:
Device: Lens A — daily disposable soft contact lens - test lens
Device: Lens B — daily disposable soft contact lens - control lens

SUMMARY:
The objective of the study is to compare the clinical performance of two different daily disposable, SiHy toric contact lens types, Lens A and Lens B, in existing soft lens wearers when worn for one week each.

DETAILED DESCRIPTION:
This study is a prospective, bilateral eye, double-masked, randomized, 1-week cross-over, daily-wear design involving two different daily disposable toric lens types. Each lens type will be worn for approximately one week, during which participants record their subjective lens-wear experience.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Self reports having a full eye examination in the previous two years;
* Anticipates being able to wear the study lenses for at least 12 hours a day, 7 days a week;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Habitually wears toric soft contact lenses binocularly, of any replacement frequency, for the past 3 months minimum;
* Has refractive astigmatism at least -0.75DC in each eye, maximum -2.25DC;
* Has refractive cylinder axis either between 155 to 25 or between 65 and 115 degrees;
* Is myopic and requires a spectacle spherical component of -1.00D to -6.50D inclusively;
* Can be fit and achieve binocular distance vision of at least 20/30 Snellen with the available lens parameters

Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Habitually wears one of the study contact lenses;
* Has any known active ocular disease and/or infection that contraindicates contact lens wear;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
* Has known sensitivity to the diagnostic sodium fluorescein used in the study;
* Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
* Has undergone refractive error surgery or intraocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Study Director — Centre for Ocular Research and Education
Locations (4):
- United States (4):
  - Golden Optometric Group, Whittier, California
  - Golden Vision, Sarasota, Florida
  - Sacco Eye Group, Vestal, New York
  - Athens Eye Care, Athens, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens A, Then Lens B: Subjects will be randomized to wear test lenses for one week and then cross-over to control lenses for one week.
  Lens A: daily disposable soft contact lens - test lens
  Lens B: daily disposable soft contact lens - control lens
- Lens B, Then Lens A: Subjects will be randomized to wear control lenses for one week and then cross-over to test lenses for one week.
  Lens A: daily disposable soft contact lens - test lens
  Lens B: daily disposable soft contact lens - control lens
Period: First Intervention
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 24 | 24
Completed | 24 | 23
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 24 | 23
Completed | 24 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: daily disposable soft contact lens - test lens
  Subjects will be randomized to wear test lenses for one week and then cross-over to control lenses for one week.
  Lens A: daily disposable soft contact lens - test lens
  Lens B: daily disposable soft contact lens - control lens
Arm/Group | Overall Study
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Ease of Lens Handling
Description: Ease of overall lens handling for putting on eyes, removing from eyes, and opening packaging will be measured on a 0-10 integer scale (0=Very difficult, 10-Very easy)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lens A: Subjects will be randomized to wear test lenses for one week and then cross-over to control lenses for one week.
  Lens A: daily disposable soft contact lens - test lens
- Lens B: Subjects will be randomized to wear control lenses for one week and then cross-over to test lenses for one week.
  Lens B: daily disposable soft contact lens - control lens
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 47 | 47
units on a scale | 9.0 (1.1) | 8.8 (1.5)

2. Secondary Outcome: Visual Acuity
Description: Visual acuity will be measured using LogMAR scale in high room illumination high contrast: distance (≥4m)
Time Frame: Baseline - after lenses have settled for 10 minutes
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 47 | 47
logMAR | -0.06 (0.06) | -0.06 (0.06)

3. Secondary Outcome: Visual Acuity
Description: Visual acuity will be measured using LogMAR scale in high room illumination high contrast: distance (≥4m)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 47 | 47
logMAR | -0.06 (0.06) | -0.05 (0.06)

ADVERSE EVENTS:
Time Frame: From dispense up to 1 week on each study lenses for a total of 2 weeks
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 1/48
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens A (N=48) | Lens B (N=48)
inferior single corneal peripheral ulcer (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT04831515/Prot_SAP_000.pdf